CLINICAL TRIAL: NCT07200999
Title: Prevalence of Carriage of Extended-Spectrum Beta-Lactamase (ESBL)-Producing Enterobacteria in Preterm Premature Rupture of Membranes : A French Multicenter Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0117_SMIT
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: Premature Rupture of Membranes; Enterobacteriaceae; Beta-Lactams; Drug Resistance, Bacterial; Antibiotic Prophylaxis; Pregnancy; Intrauterine Infection
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at how common certain antibiotic-resistant bacteria (called extended-spectrum beta-lactamase-producing Enterobacteriaceae, or E-BLSE) are in pregnant women who experience premature breaking of their water before full term. The goal is to understand how often these bacteria are found, how long they stay, and what factors increase the risk of carrying them. This information will help doctors choose the best antibiotics to protect both the mother and baby from infections during and after pregnancy. The study follows women from the time of their membrane rupture until delivery, collecting samples to track the bacteria over time.

ELIGIBILITY:
Inclusion Criteria :

* Pregnant women aged over 18 years
* Diagnosed with premature rupture of membranes before term (between 23 weeks + 0 days and 36 weeks + 6 days of gestation)
* Managed in one of the participating maternity hospitals

Exclusion Criteria :

* No available microbiological sample
* Minors or women under legal guardianship (curatorship, tutelage, or judicial protection)
* Women who refuse the use of their clinical data for research purposes at admission or within one month after receiving the information document

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study participants will be selected from pregnant women who experience premature rupture of membranes before term (between 23 weeks and 36 weeks + 6 days of gestation). These women will be receiving care at multiple maternity hospitals participating in this multicenter French study. The population includes adult women (over 18 years old) who have vaginal microbiological samples available for analysis. This group represents a high-risk pregnancy population due to the increased risk of infection associated with premature membrane rupture.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
The proportion of vaginal swabs (PV) positive for extended-spectrum beta-lactamase-producing Enterobacteriaceae (E-BLSE) in pregnant women with premature rupture of membranes before term, measured at diagnosis, during the latency period, and at delivery. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Denis, Saint-Denis, France, France